CLINICAL TRIAL: NCT03708601
Title: Prognostic Risk of Patients With Essential Hypertension for Cardiovascular Events
Brief Title: Prognostic Risk of Patients With Essential Hypertension for Cardiovascular Events (PROSPECT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Shanxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PROSPECT
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2018-06

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry study aims to determine serial biomarkers to prognosis of Essential Hypertension

DETAILED DESCRIPTION:
The study aims to investigate the role of candidate biomarkers in the prognosis of Essential Hypertension. In the prognosis part of the study, patients with confirmed hypertension are enrolled. The outcome is unstable angina, coronary revascularization, acute myocardial infarction, heart failure, atrial fibrillation, ischemic cerebral infarction, hemorrhagic cerebral infarction, transient ischemic attack, doubling of serum creatinine or end-stage renal disease (defi ned as eGFR less than 15 mL/min/1·73 m² or need for chronic dialysis) and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the study program were as follows:

Men or women of any racial background, 18 years of age and older, with systolic BP greater than or equal to160 mm Hg, and presence of three or more cardiovascular risk factors or disease.

The qualifying risk factors were male sex, age older than 50 years, verified diabetes mellitus, current smoking, high total cholesterol, left ventricular hypertrophy by electrocardiogram, proteinuria on dipstick and raised serum creatinine between 150 and 265 umol/L. The qualifying diseases were verified coronary disease, cerebrovascular disease or peripheral arterial occlusive disease, or left ventricular hypertrophy with strain pattern.

Exclusion Criteria:

The exclusion Criteria for the study program were as follows:

Secondary hypertension, pregnancy, history of heart failure or left ventricular ejection fraction less than 40%, myocardial infarction within one month, percutaneous transluminal coronary angioplasty or coronary artery bypass grafting, cerebrovascular disease, severe liver disease, severe chronic renal failure (eGFR less than 30 mL/min/1.73 m2) in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The case group consists of patients who was diagnosed as Essential Hypertension; control group is general population without Essential Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-09-08 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-08-08 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular adverse events | These data is collected from the cases' medical record or during follow-up visit at 1-3 years after discharge.
  Number of cardiovascular adverse events including unstable angina, coronary revascularization, acute myocardial infarction, heart failure, atrial fibrillation. revascularization, myocardial infarction, heart failure
Number of cerebrovascular adverse events | These data is collected from the cases' medical record or during follow-up visit at 1-3 years after discharge.
  Number of cerebrovascular adverse events including ischemic stroke and hemorrhagic stroke.
Number of renal adverse events | These data is collected from the cases' medical record or during follow-up visit at 1-3 years after discharge.
  Number of renal adverse events including Double serum creatinine or end-stage renal disease (eGFR less than 15 mL/min/1.73 m2 or dialysis required).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PhD, Study Director — The Key Laboratory of Remodeling-Related Cardiovascular Disease, Ministry of Education, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart,Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yin W, Li F, Tan X, Wang H, Jiang W, Wang X, Li S, Zhang Y, Han Q, Wang Y, Du J. Plasma Ceramides and Cardiovascular Events in Hypertensive Patients at High Cardiovascular Risk. Am J Hypertens. 2021 Nov 20;34(11):1209-1216. doi: 10.1093/ajh/hpab105. PMID 34232291